CLINICAL TRIAL: NCT04833946
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess the Effect of 336 Days Exposure of Paractin® on Pain & Disease Progression in Patients Suffering From Osteoarthritis of Knee Joint.
Brief Title: To Assess the Effect of 336 Days Exposure of Paractin® on Pain & Disease Progression in Patients Suffering From Osteoarthritis of Knee Joint.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IN/201001/PARACTIN/OA
Record Dates: First submitted 2021-04-03; First posted 2021-04-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis (Knee OA)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Andrographis paniculata extract; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Andrographis paniculata [150 mg] (Active Comparator): One capsule to be taken orally, 30 minutes after breakfast & 30 minutes before bedtime
  Interventions: Other: Andrographis paniculata [150 mg]
- Microcrystalline Cellulose (MCC) (Placebo Comparator): One capsule to be taken orally, 30 minutes after breakfast & 30 minutes before bedtime
  Interventions: Other: Microcrystalline Cellulose (MCC)

INTERVENTIONS:
Other: Andrographis paniculata [150 mg] — One capsule to be taken orally, 30 minutes after breakfast & 30 minutes before bedtime
  Arms: Andrographis paniculata [150 mg]
Other: Microcrystalline Cellulose (MCC) — One capsule to be taken orally, 30 minutes after breakfast & 30 minutes before bedtime
  Arms: Microcrystalline Cellulose (MCC)

SUMMARY:
Sponsor aimed to study hydroalcoholic extract of Andrographis paniculata (for its effect on OA disease progression in OA patients with moderate to severe knee OA.

Hydroalcoholic extract of Andrographis paniculata (standardized for 50% bioactive andrographolides).Andrographis paniculata may have an effect on increasing the expression of collagen type II protein and also mitigate the migration of inflammatory cells or angiogenesis

DETAILED DESCRIPTION:
Sponsor aimed to study hydroalcoholic extract of Andrographis paniculata (for its effect on OA disease progression in OA patients with moderate to severe knee OA.

Hydroalcoholic extract of Andrographis paniculata (standardized for 50% bioactive andrographolides). It has been evaluated in clinical studies for its anti-inflammatory and anti-oxidant activities. Although the potential cartilage regenerative mechanism of Andrographis paniculata is unknown, Sponsor believe that Andrographis paniculata may have an effect on increasing the expression of collagen type II protein and also mitigate the migration of inflammatory cells or angiogenesis. In the present study, knee morphometrics (joint space narrowing of tibiofemoral joint, and cartilage thickness at the femur, tibia and patella compartments), cartilage turnover (serum COMP levels), bone turnover (serum Bone specific alkaline phosphatase) along with symptomatic relief (Using mWOMAC) in patients with primary knee OA over a period of 336 days will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female Patients aged ≥40 and ≤85 years.
2. Patients with a history of clinically symptomatic OA of the knee for ≥ 6 months.
3. Index knee joint pain rated ≥60 mm on a 100 point Pain Visual Analogue Scale (VAS).
4. Patient must have a diagnosis of idiopathic OA according to the American College of Rheumatology clinical and radiographic criteria with knee pain, osteophytes, and fulfilment of at least 2 of the 3 criteria:

   * Age of ≥50 years Stiffness lasting <30 minutes after getting up in the morning
   * Crepitus
5. Radiographic evidence of grade II- III knee OA based on the Kellgren and Lawrence (KL) radiographic entry criteria for OA.

   * Grade II: - Definite osteophytes and possible joint space narrowing (JSN) on the anteroposterior weight-bearing radiograph.
   * Grade III: Anteroposterior weight-bearing knee radiograph demonstrates definite joint space narrowing, multiple osteophyte formations, some sclerosis, and possible deformity of bony ends.
6. Patients with normal liver & renal function defined as:

   * Serum Alkaline phosphatase levels up to 1.5 of ULN (Upper Limit of Normal).
   * Serum AST and ALT levels up to 2.5 of ULN.
   * Serum creatinine levels up to 1.5 of ULN.
   * Blood Urea Nitrogen levels up to 1.5 of ULN.
7. Female Patients must not be of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy])
8. Patients must be willing to discontinue any NSAIDs or other analgesic (eg, aspirin, acetaminophen) or potentially confounding concomitant treatments (eg, physiotherapy, acupuncture) starting from the screening visit until completing participation in the study.
9. Abstinence from any home-based remedies or any other form of topical products intended for knee joint pain relief for the entire study duration.
10. Patient must be willing to avoid unaccustomed physical activity (eg, starting a new weight lifting routine) for the duration of the study starting from the screening visit.
11. Ability to read and provide written, personally signed, and dated informed consent to participate in the study.
12. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. Patients who have any contraindications to MRI, such as, but not limit to:A metal device affected by MRI (e.g. any type of electronic, mechanical, or magnetic implant; cardiac pacemaker; aneurysm clip(s); implanted cardiac defibrillator); - Have history of orbit trauma by a potential ferromagnetic foreign body (metal slivers, metal shavings, other metal objects) for which they sought medical attention; - Have claustrophobia; - Have difficulty fitting into the MRI knee coil due to greater than normal thigh diameter.
2. Any other lower limb dis-functionality of lower limb other than the knee that, in the opinion of the Investigator, could interfere with pain and functional assessments related to the knee.
3. Patients who has a history of total or partial knee replacement, arthroplasty, or other knee surgery on either knee.
4. Patients who has had significant injury, as judged by the Investigator, involving the target knee within the 6 months before screening.
5. Patients who has used opiates or corticosteroids within 30 days before screening for the target knee or who requires treatment with chronic opiates or corticosteroids or had intra articular injections of corticosteroids, hyaluronic acid, or visco supplements to a knee to be treated within the 3 months before Screening.
6. Patients who has a history of significant hypersensitivity, intolerance, or allergy to ibuprofen, any NSAIDs, aspirin, or acetaminophen.
7. Known sensitivity to the investigational product or any excipients of the drug product.
8. Patients who has a history of chronic inflammatory disease (such as rheumatoid arthritis, psoriatic arthritis, gouty arthritis), fibromyalgia, or other conditions that may affect the target joint or the functional and pain assessments (eg, osteonecrosis, chondrocalcinosis).
9. Patients has any clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease, or any other condition that, in the investigator's opinion, could compromise the Patient's welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.
10. Patients has any other clinically significant laboratory finding at screening that in the investigator's opinion contraindicates study participation.
11. Presence of uncontrolled hypertension (Defined as SBP ≥ 140 mm Hg and/or DBP ≥ 90 mm Hg).
12. Uncontrolled diabetes defined as fasting blood glucose (FBG) > 125 mg/dL.
13. Patients with heavy alcohol consumption, defined as - For men: More than 14 standard alcoholic drink (SAD)/week or more than 4 SAD in a day. - For women: More than 7 SAD/week or more than 3 SAD in a day.

    (NOTE - A standard alcoholic drink contains approximately 14 grams of alcohol, which is equivalent to 12 ounces of beer (~5% alcohol), 8.5 ounces of malt liquor (~9% alcohol), 5 ounces of wine (~12% alcohol), 3.5 ounces of fortified wine (e.g., sherry or port), or 1.5 ounces of liquor (distilled spirits; ~40% alcohol).
14. Binge drinkers, defined as 4 or more SAD for women, and 5 or more SAD for men, in a 2-hour time frame.
15. Individuals having a history (in past 2 years) of smoking or currently smoking or using any form of smokeless tobacco.
16. Patients without access to telephone and/or ability to gain technology access.
17. Patients who participated in another human trial within last 90 days prior to screening.
18. Any condition that could, in the opinion of the investigator, preclude the Patient's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Joint Space Narrowing as assessed by magnetic resonance imaging | Day 0 and day 336
  to evaluate the effect of 336 days of IP consumption on change in joint space narrowing (JSN) in the tibiofemoral joint of knee as measured by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Modified Western Ontario and McMaster Universities Pain and total scores | day 0, 28, 84, 140, 168, 252 and day 336
  Patients rate their pain, stiffness, or physical function using five ordinal responses: none, mild, moderate, severe, and extreme..Change in knee joint pain as assessed by the Western Ontario and McMaster University Arthritis Index pain subscale (mWOMAC -P)
Cartilage thickness at femur, tibia and patella compartments | Day 0 and day 336
  Change in cartilage thickness at the femur, tibia and patella compartments as assessed by MRI
Outcome Measures in Arthritis Clinical Trials OA Research Society International | day 336
  Treatment responders as assessed by OMERACT-OARSI in comparison to placebo
Bone turnover (by measuring bone specific alkaline phosphatase levels) | Day 0 and day 336
  Change in bone turnover as assessed by change in serum levels of bone specific alkaline phosphatase
Cartilage turnover as assessed by Cartilage Oligomeric matrix protein (COMP) | Day 0 and day 336
  Change in cartilage turnover as assessed by change in serum levels of cartilage oligomeric matrix protein
Change in the Quality of Life | Day 0, 84, 168, and day 336
  Change in Quality of life as assessed by using Short Form-36

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - Ayush Nursing Home, Mumbai, Maharashtra
  - New Healthcare Nursing Home, Thane, Maharashtra
  - Jaipur National University Institute for Medical Sciences and Research Center, Jaipur, Rajasthan
  - Asopa Hospital, Jaipur, Rajasthan
  - Shubham Sudbhawana Super Specialty Hospital, Varanasi, Uttar Pradesh